CLINICAL TRIAL: NCT04937075
Title: Impact of Antimicrobial Stewardship on Outcomes of Patients With Hospital-acquired Pneumonia Due to Gram-negative Bacilli - A Before-after ORACLE Study
Brief Title: Impact of Antimicrobial Stewardship on Outcomes of Patients With Hospital-acquired Pneumonia Due to Gram-negative Bacilli - A Before-after Study
Acronym: ORACLE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0066
Record Dates: First submitted 2021-05-31; First posted 2021-06-23 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: Hospital-acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before period without multiplex PCR identification
  Interventions: Other: No intervention
- After period with multiplex PCR identification
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Hospital-acquired pneumonia (HAP) is one of the most frequent complications and the main cause of antibiotics use in hospitalized patients, particularly in intensive care units (ICUs). The latest European and French recommendations for the management of HAP were published in 2017 and 2018. Gram-negative bacilli are frequently identified in this pneumonia.

The experts discussed the issue of tailored-empiric antimicrobial therapy. Because delayed antimicrobial therapy is associated with poor outcomes, their conclusion was to reduce the time to deliver proper antimicrobial therapy, but to limit over-use of broad-spectrum molecules. Since delays in microbiological identification hinder the ability of clinicians to streamline therapy, rapid diagnostic with multiplex PCR, which decreases the time to organism identification by 2 days compared to conventional methods, is appealing, especially for gram-negative bacilli. The FilmArray® Lower Respiratory Tract Infection Panel is a rapid multiplex PCR which tests for the most frequently pathogens (18 bacteria including plenty of gram-negative bacilli +5 genes of resistance, and 9 viruses) involved in HAP. The FilmArray® Lower Respiratory Tract Infection (LRTI) Panel has a sensitivity and a specificity of 95% and 99% respectively and can be implemented in a personalized antimicrobial guidance to treat HAP due to gram-negative bacilli. The investigators hypothesized that a rapid multiplex PCR for guidance of empiric antimicrobial therapy, especially for gram-negative bacilli, reduces the time-to-proper antimicrobial therapy and reduces the risk of death of patients suffering of HAP.

The investigators aim to assess the efficacy of an antimicrobial stewardship including the results of a rapid respiratory panel multiplex PCR for empiric antimicrobial guidance in patients with hospital-acquired pneumonia due to gram-negative bacilli.

The investigators will use a before-after design to test the efficiency of an antimicrobial stewardship including a highly innovative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent adult patients
* Receiving mechanical ventilation
* Suspected hospital-acquired pneumonia
* Non-opposition from the patient or a relative.

Exclusion Criteria:

* Pregnant women, breastfeeding-women
* Minors, Adults under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include 400 patients hospitalized in intensive care units, under mechanical ventilation, with a suspected hospital-acquired pneumonia : 200 patients in the retrospective "before" phase, 200 patients in the prospective "after" phase with the PCR multiplex identification
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of access to empiric antibiotic therapy guided by Multiplex PCR in intensive care patients with hospital acquired pneumonia | 28 days
  Composite endpoints: survival on D28, number of days without mechanical ventilation on D28, and clinical recovery between D7 and D10 (RADAR method)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nantes, Nantes
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: Undecided